CLINICAL TRIAL: NCT01980355
Title: The Effect of Tranexamic Acid on Blood Loss and Transfusion Rates in Major Oncologic Surgery
Brief Title: TXA Study in Major Oncologic Surgery
Acronym: TXA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health West (Other)
Responsible Party: Principal Investigator, Gerald P. Wright, Surgical Oncology and Hepatopancreaticobiliary Surgeon, Corewell Health West
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-133
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Results first posted 2022-05-05 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Tranexamic Acid; Cancer; Major Surgery
Keywords: cancer; surgery; oncology; major; surgical oncology; tranexamic acid
MeSH Terms: conditions — Neoplasms | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic Acid (Experimental): 1000mg tranexamic acid; given over 15 minutes into the vein once prior to surgery.
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): Placebo given over 15 minutes into the vein once prior to surgery.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid
  Arms: Tranexamic Acid
Other: Placebo
  Arms: Placebo

SUMMARY:
Major surgery can result in blood loss that can require a blood transfusion during and/or after surgery. Tranexamic acid is a medication that was first introduced in the 1960s as a treatment for heavy menstrual bleeding. Over the past 20 years it has been used and studied in patients undergoing open-heart surgery, liver transplantation, and urologic surgery. We believe tranexamic acid may possibly decrease bleeding related to major surgery, resulting in reduced blood loss, lower blood transfusion rates, and possibly decreased hospital costs related to your surgical hospital stay.

In this study, you will receive either the drug tranexamic acid or a placebo. The placebo looks like the tranexamic acid, but does not have any active ingredient in it. The treatment you get will be chosen by chance, like flipping a coin. You will have equal chance of being given the tranexamic acid or the placebo. In this study, both the tranexamic acid and the placebo are considered research.

DETAILED DESCRIPTION:
Neither you nor the study doctor will choose what treatment you get. You will have an equal chance of being given the tranexamic acid or the placebo. Neither you nor the study doctor will know which treatment you are getting.

You will receive one 1000 mg dose of either tranexamic acid or placebo immediately before surgery. This dose of tranexamic acid or placebo will be given in your vein over 15 minutes.

Information from your medical record related to your surgery and recovery time in the hospital will be collected by medical staff assisting with this study and recorded on study forms. These study forms will be labeled with your study number instead of your name. Additionally, if you return to the hospital within 90 days after you went home from the hospital, information about that hospital visit(s) will also be collected from your medical record.

ELIGIBILITY:
Inclusion Criteria

* Subjects undergoing major oncologic surgery for standard of care purposes (to include, but not limited to: liver resections, radical cholecystectomy, pancreaticoduodenectomy (Whipple procedure), esophagectomy, gastrectomy, colectomy, debulking with hyperthermic intraperitoneal chemotherapy, prostatectomies, nephrectomies and partial nephrectomies)
* Male or female > 18 years of age
* Subject agrees to participate in this study and provides informed consent

Exclusion Criteria

* Subjects with a history of hypercoagulopathy, deep vein thrombosis or pulmonary embolism
* Subjects that are on therapeutic anticoagulation or therapeutic antiplatelet medications at the time of surgery other than Aspirin
* Subjects with a history of TIA or stroke
* Subjects with a history of atrial fibrillation
* Subjects with a known thrombus
* Baseline creatinine level greater than 2.83 mg/dL
* Subjects with known hypersensitivity to tranexamic acid
* Adults unable to provide informed consent
* Children
* Pregnant women
* Prisoners
* Non-English speaking subjects
* Any other medical condition including mental illness or substance abuse deemed by the investigator to be likely to interfere with a subject's ability to provide informed consent, cooperate and take part in this research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-06-12 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2020-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald P Wright, MD, Principal Investigator — Corewell Health West
Locations (1):
- Spectrum Health Hospitals, Grand Rapids, Michigan, United States

REFERENCES:
- [Background] Vermylen J, Verhaegen-Declercq ML, Verstraete M, Fierens F. A double blind study of the effect of tranexamic acid in essential menorrhagia. Thromb Diath Haemorrh. 1968 Dec 31;20(3):583-7. No abstract available. PMID 5710474
- [Background] Casati V, Gerli C, Franco A, Torri G, D'Angelo A, Benussi S, Alfieri O. Tranexamic acid in off-pump coronary surgery: a preliminary, randomized, double-blind, placebo-controlled study. Ann Thorac Surg. 2001 Aug;72(2):470-5. doi: 10.1016/s0003-4975(01)02802-8. PMID 11515884
- [Background] Massicotte L, Denault AY, Beaulieu D, Thibeault L, Hevesi Z, Roy A. Aprotinin versus tranexamic acid during liver transplantation: impact on blood product requirements and survival. Transplantation. 2011 Jun 15;91(11):1273-8. doi: 10.1097/TP.0b013e31821ab9f8. PMID 21617589
- [Background] Crescenti A, Borghi G, Bignami E, Bertarelli G, Landoni G, Casiraghi GM, Briganti A, Montorsi F, Rigatti P, Zangrillo A. Intraoperative use of tranexamic acid to reduce transfusion rate in patients undergoing radical retropubic prostatectomy: double blind, randomised, placebo controlled trial. BMJ. 2011 Oct 19;343:d5701. doi: 10.1136/bmj.d5701. PMID 22012809
- [Background] CRASH-2 trial collaborators; Shakur H, Roberts I, Bautista R, Caballero J, Coats T, Dewan Y, El-Sayed H, Gogichaishvili T, Gupta S, Herrera J, Hunt B, Iribhogbe P, Izurieta M, Khamis H, Komolafe E, Marrero MA, Mejia-Mantilla J, Miranda J, Morales C, Olaomi O, Olldashi F, Perel P, Peto R, Ramana PV, Ravi RR, Yutthakasemsunt S. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2): a randomised, placebo-controlled trial. Lancet. 2010 Jul 3;376(9734):23-32. doi: 10.1016/S0140-6736(10)60835-5. Epub 2010 Jun 14. PMID 20554319
- [Background] Cap AP, Baer DG, Orman JA, Aden J, Ryan K, Blackbourne LH. Tranexamic acid for trauma patients: a critical review of the literature. J Trauma. 2011 Jul;71(1 Suppl):S9-14. doi: 10.1097/TA.0b013e31822114af. PMID 21795884
- [Background] Wu CC, Ho WM, Cheng SB, Yeh DC, Wen MC, Liu TJ, P'eng FK. Perioperative parenteral tranexamic acid in liver tumor resection: a prospective randomized trial toward a "blood transfusion"-free hepatectomy. Ann Surg. 2006 Feb;243(2):173-80. doi: 10.1097/01.sla.0000197561.70972.73. PMID 16432349
- [Background] Kalavrouziotis D, Voisine P, Mohammadi S, Dionne S, Dagenais F. High-dose tranexamic acid is an independent predictor of early seizure after cardiopulmonary bypass. Ann Thorac Surg. 2012 Jan;93(1):148-54. doi: 10.1016/j.athoracsur.2011.07.085. Epub 2011 Nov 4. PMID 22054656
- [Background] Henry DA, Carless PA, Moxey AJ, O'Connell D, Stokes BJ, McClelland B, Laupacis A, Fergusson D. Anti-fibrinolytic use for minimising perioperative allogeneic blood transfusion. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD001886. doi: 10.1002/14651858.CD001886.pub2. PMID 17943760

RESULTS

PARTICIPANT FLOW:
Groups:
- Tranexamic Acid: 1000mg tranexamic acid; given over 15 minutes into the vein once prior to surgery.
  Tranexamic Acid
- Placebo: Placebo given over 15 minutes into the vein once prior to surgery.
  Placebo
Period: Overall Study
Arm/Group | Tranexamic Acid | Placebo
Started | 39 | 37
Completed | 39 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid | Placebo | Total
Number analyzed (Participants) | 39 | 37 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (11.9) | 63.2 (11.2) | 61.1 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 29 | 30 | 59
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Required Transfusion
Description: To determine the impact of perioperative administration of tranexamic acid on blood loss and transfusion rates in major oncologic surgery
Time Frame: From time of surgery to 90 days post hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 39 | 37
Participants | 8 | 5

2. Secondary Outcome: Estimated Blood Loss
Description: Surgical blood loss estimation
Time Frame: From time of surgery to 90 days post hospital discharge
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 39 | 37
mL | 450 [250 to 750] | 365 [150 to 850]

ADVERSE EVENTS:
Time Frame: 90 days from the time of surgery
Description: Morbidity graded according to Clavien-Dindo classification
Arm/Group | Tranexamic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 2/39 | 0/37
Serious Adverse Events (participants affected / at risk) | 11/39 | 13/37
Other Adverse Events (participants affected / at risk) | 0/39 | 0/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tranexamic Acid (N=39) | Placebo (N=37)
Surgical Morbidity (Surgical and medical procedures) | 11 (11) | 13 (13) — Clavien-Dindo Grade III or higher

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-11-20): https://cdn.clinicaltrials.gov/large-docs/55/NCT01980355/Prot_SAP_000.pdf
  • Informed Consent Form (2017-09-19): https://cdn.clinicaltrials.gov/large-docs/55/NCT01980355/ICF_001.pdf